CLINICAL TRIAL: NCT04884659
Title: The Impact of Time-Restricted Feeding on Metabolism and Inflammation in Obesity (TRIO Study)
Brief Title: Time-Restricted Feeding
Acronym: TRIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JAL-1007
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Inflammatory Markers; Glycemic Variation; Time Restricted Feeding; Ketosis
MeSH Terms: conditions — Obesity; Intermittent Fasting; Ketosis

STUDY DESIGN:
Intervention Model Description: 10 obese, pre-diabetic participants will be randomly assigned to usual eating pattern vs timed restricted eating over 5 days as inpatient in a metabolic unit. They will undergo baseline and post-intervention measurements of glucose tolerance, body compostion by Bod Pod, continuous glucose monitoring by Free-Syle Libre monitor and donate blood for markers of inflammation. They will consume their usual pre-study diet. After completing Arm I, they will cross-over to Arm 2.
Who Masked: Participant, Investigator
Masking Description: Investigator and participants will be blinded to randomization prior to initiation of study arm. The randomization will be determined by the research pharmacist. Since the arms require different timing of meals it will be obvious as to the arm, once it is started. However, neither the investigator nor the participant can choose the order of the arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Timed restricted feeding (Experimental): Time restricted feeding then usual feeding pattern Day 1, testing
  Day 2-7 all meals will be consumed as follows:
  80% of calories consumed before 2 PM with remaining 20% consumed by 4PM. Fasting except for water, non caloric drinks for 14-16 hours Same number of calories consumed as in usual feeding pattern arm. Day 8 testing. Day 9-14 crossover to usual feeding pattern arm (meals consumed ad lib with 50% of calories consumed after 4 PM) for 6 days.
  Interventions: Other: Time restricted feeding arm; Other: usual feeding pattern arm
- Usual feeding pattern (Experimental): Usual feeding pattern, then time restricted feeding Day 1 testing
  Day 2-7 all meals will be consumed as follows:
  Meals consumed ad lib with 50% of calories consumed after 4 PM. Day 8 testing. Day 9-14 crossover to time restricted feeding arm with all meals consumed as follows:
  80% of calories consumed before 2 PM with remaining 20% consumed by 4PM. Fasting except for water, non caloric drinks for 14-16 hours Same number of calories consumed as in usual feeding pattern arm for 6 days.
  Interventions: Other: Time restricted feeding arm; Other: usual feeding pattern arm

INTERVENTIONS:
Other: Time restricted feeding arm — 80% of calories consumed before 2PM, remaining 20% consumed by 4PM. Fasting for 14-16 hours
Other: usual feeding pattern arm — All meals consumed ad lib with 50% of calories consumed after 4PM

SUMMARY:
We propose to conduct a randomized 6-day isocaloric crossover feeding study in humans with prediabetes and obesity. We will study the effect of restricting the timing of caloric intake to earlier in the day (TRF) versus later in the day (usual feeding pattern, UFP) on glycemia and inflammation in an inpatient setting.

DETAILED DESCRIPTION:
Time Restricted Feeding (TRF) is a variant of intermittent fasting that confines caloric intake to active daytime hours and involves fasting for 12 to 14 hours. Circadian misalignment caused by changes in sleeping and eating behaviors has emerged as having a detrimental impact on weight, glucose homeostasis and other cardiovascular disease-related outcomes. Feeding during active periods appears to be advantageous for weight, glucose metabolism and lipid profiles whereas feeding during the inactive period confers deleterious effects on these outcomes. Therefore, TRF shows great promise as a novel intervention for addressing obesity and related cardiovascular outcomes.

Animal studies suggest that timing of feeding, including intermittent fasting or TRF, decreases inflammation and causes ketosis. Human studies that examined time restricted feeding for improvement in glycemia in as little as 4 days did not observe changes in clinical markers of inflammarion such as hsCRP. Moreover, systemic and adipose tissue inflammation as it occurs in obesity shows dynamic changes in the context of weight loss that would not be clearly apparent in a weight stable state. A potential mechanistic link between glycemic improvement and systemic inflammation would be the Receptor for Advanced Glycation End-Products (RAGE) and its soluble form (sRAGE).This form of inflammation has not been measured in reported eTRF studies and its relationship with eTRFwould bea significant contribution from the proposed study.

ELIGIBILITY:
Inclusion Criteria:

1. BMI >25 kg/m2
2. If taking probiotics during screening, must agree to continue taking them at the same dosage and frequency
3. HbA1C 5.7-6.4%
4. Willing to eat only the food provided
5. Willing to follow the feeding schedule, including fasting for 14 hours/day for 7 days
6. Willing to remain on the RU inpatient 24/7 unit except for weekend passes
7. Normally sleep between the hours of 10 pm and 8 am
8. Weight stable over the last 3 months defined as no more than a 5% change

Exclusion Criteria:

1. Diabetes
2. Any intermittent feeding diet within the last 2 weeks
3. HIV positive
4. Hepatitis
5. Self-reported autoimmune diseases (rheumatoid arthritis, SLE (lupus), Crohn's
6. Disease, psoriasis, etc.)
7. Current use of metformin
8. Smoked tobacco within the last 8 weeks
9. Taking any weight loss medication
10. Current use of systemic steroids
11. Allergic to adhesive tape
12. Taking clinically useful medications that contribute to significant weight loss or weight gain ie tricyclic antidepressants, some SSRIs, lithium, antipsychotics, some anticonvulsants, steroids, beta blockers, some antihistamines.
13. Currently pregnant
14. Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Change in glycemic variation by mean amplitude of glycemic excursion (MAGE) | Day 2-Day14
Change in inflammatory marker concentrations (sRAGE and hsCRP) relative to the UFP arm | Day 2-Day 14

SECONDARY OUTCOMES:
Shift from glucogenic to ketogenic metabolism in the TRF arm relative to the UFP arm by plasma metabolomics | Day 2- Day 14
Change in biological indices of appetite (incretins) in TRF arm relative to UFP arm. | Day 2 - Day 14
Changes in WBC transcriptomic profiles versus UFP arm between1, 7 and 14 days. | Day 2 - Day 14
changes in gut mirobiome profiles in the TRFarm | Day 2 - Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- The Rockefeller University Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No